## **COVER PAGE OF STATISTICAL ANALYSIS PLAN**

Study title: Prospective Observational Study of the

PowerPICC Family of Devices and

Accessories

Protocol number.: MDS-19PICCEU01

NCT number: **NCT04263649** 

Statistical Analysis Plan v.5.0, 28-March 2022

version and date:



# Statistical Analysis Plan for interim and final analysis

#### Version 5.0

Study: Prospective Observational Study of the Power PICC Family of Devices and

Accessories

Study-ID: MDS-19PICCEU01

Sponsor / Contact: Becton Dickinson and Company

Bard Access Systems 605 North 5600 West Salt Lake City, Utah 84116

**United States** 

Evaluation: FGK Clinical Research GmbH

FGK code 3558

Version: 5.0 of 28Mar2022 (final)

Previous versions: 4.0 of 28Jul2021 (final)

3.0 of 16Apr2021 (final) 2.0 of 15Apr2021 (final) 1.0 of 23Dec2020 (final)

The content of this Statistical Analysis Plan is confidential and must not be passed to any third party without permission of Becton Dickinson and Company.



## **Revision history**

| Version | Author | Date | Reason for Revision |
|---|---|---|---|
| 2.0 | P. Wolf | 15Apr2021 | Derivation of performance success clarified; title used for all generated TLGs adapted; appendix updated |
| 3.0 | P. Wolf | 16Apr2021 | Assignment of analysis sets to analysis adapted |
| 4.0 | P. Wolf | 28Jul2021 | Section 4.4.2: derivation of incidence of complications adapted (only non-missing values used for calculation of percentages) Section 4.4.3: MedDRA version 23.0 added Section 5 added |
| 5.0 | P. Wolf | 28Mar2022 | <ul> <li>Analysis of safety and performance endpoints adapted to only use non-missing values for the calculation of percentages.</li> <li>Ease of insertion questionnaire: exception added that specific missing values will be set to not applicable/ not used</li> </ul> |



#### **Table of Contents**

| RE' | VISION H | 1ISTORY | 2 |
|---|---|---|---|
| TAI | BLE OF | CONTENTS | 3 |
| LIS | T OF AB | BREVIATIONS | 4 |
| 1 | GENER | AL | 5 |
| • | 1.1<br>1.2<br>1.3<br>1.4 | Overall Design | 6<br>6 |
| 2 | SAFET | Y AND PERFORMANCE VARIABLES | 7 |
| | 2.1<br>2.2<br>2.3<br>2.4<br>2.5 | Primary Safety Variable | 7<br>7 |
| 3 | STATIS | TICAL ANALYSIS SETS | 8 |
| | 3.1<br>3.2<br>3.3<br>3.4<br>3.5 | Enrolled Set Safety Set Evaluable Set Additional Subgroup Analysis Assignment of Analysis Sets to Analysis | 8<br>8 |
| 4 | STATIS | TICAL EVALUATION | 9 |
| | 4.1<br>4.2<br>4.3<br>4.4<br>4.4.1<br>4.4.2<br>4.4.3 | Dispositions of Participants and Analysis Sets Demographics and Other Covariates Catheter insertion, Maintenance and Removal. Safety Analysis Analysis of Primary Safety Variable Analysis of Secondary Safety Variables Further Safety Variables | 9<br>. 10<br>. 11<br>. 11 |
| | 4.5 | Performance Analysis | |
| | 4.5.1<br>4.5.2 | Analysis of Primary Performance Variable | . 12 |
| | 4.6 | Other Analysis | |
| | 4.7<br>4.8 | Missing Values | |
| | 4.0 | Data Base Closure and Data Review | |
| | 4.10 | Miscellaneous | |
| 5 | SIGNY. | TIIDES | 16 |



#### **List of Abbreviations**

In the following abbreviations are listed as used within this statistical analysis plan or which might occur within the tables, listings and graphs outputs:

AE Adverse event

BMI Body mass index

CI Confidence interval

CRF Case report form

DRM Data review meeting

EC Exclusion Criterion

IC Inclusion Criterion

ICF Informed Consent

IFU Instructions for Use

LLT Lower level term

MedDRA Medical dictionary for regulatory activities

N Number of participants

PICC Peripherally Inserted Central Catheter

PT Preferred term

SAE Serious adverse event

SAP Statistical analysis plan

SAF Safety set

SD Standard deviation

SOC System organ class

TLG Tables, listings, graphs

VT Venous Thrombosis



#### 1 General

This Statistical Analysis Plan (SAP) was defined by the Sponsor and the responsible Statistician. It is based upon the Study Protocol (version 1.0 of 12Dec2019) and contains detailed description of the statistical methods described therein.

The SAP describes prospectively the analyses to be performed on study data for the final analysis as well as for the interim analysis. It was finalized prior to the interim analysis.

#### 1.1 Overall Design

This is a prospective, observational, single arm, post-market study to assess the safety and performance of the PowerPICC family of devices. In the study, only participants who require one of the study devices may be considered for enrollment. The choice of device required for individual participants is left to the discretion of the clinician. Information will be collected on the study participants and devices before, during, and after catheter insertion, while the device is indwelling, and during device removal to assess both safety and performance. Both short- and long-term use of the PowerPICC devices will be assessed as part of the study.

#### Screening and Enrollment

After screening against inclusion/exclusion criteria, potential participants will be provided with detailed information about the study. If the potential participant, or parent/guardian in the case of those under 18 years of age, provides written informed consent, he/she will be enrolled in the study.

#### **Index Procedure**

Choice of the specific PowerPICC type, size, number of lumens, and length required for an individual patient is left to the discretion of the clinician. The device and insertion site will be prepared according to the device specific IFU. The device will be inserted, and catheter tip location will be confirmed according to standard medical practice and according to the device specific IFU. Once proper placement is confirmed, the procedure will be completed, the catheter aspirated and flushed, and secured/stabilized according to the device specific IFU. The insertion site will be dressed according to the IFU and hospital-specific protocols.

#### Use and Maintenance Procedures

The PowerPICC device will be used for therapy as medically required, according to the Instructions for Use (IFU) and hospital protocol. The device will be maintained (i.e., flushing, fluid locking, cleansing) and the site maintained (i.e., cleansing, dressing) according to the device specific IFU, standard medical practice, and hospital protocols. When the participant is treated in an acute-care setting, the catheter/site will be assessed daily until the device is removed or until they are discharged with the device in place (then treated as an outparticipant). When the participant is treated in an outparticipant setting, the catheter/site will be assessed at each therapy visit until the device is removed, or until 180 days post-insertion (±14 days), whichever comes first. For the purposes of endpoint calculations, peripherally inserted central catheters (PICCs) remaining in place after 180 days will be considered to have completed therapy.



#### **Device Removal Procedure**

The study device will be discontinued/removed when it is deemed medically appropriate by the participant's treating clinician (e.g., no longer needed, no longer functioning). Removal of the device will be performed according to the device specific IFU, standard medical practice, and hospital protocols.

#### **Investigational Sites**

Up to 20 sites in the EU will participate in this study. No more than 20% of participants may be enrolled at any one site.

#### 1.2 Sample Size Considerations

The primary safety endpoint of the study is the incidence of venous thrombosis (VT). The expected venous thrombosis rate is about 10% based on literature review. The statistical rationale of the sample size is based on precision of the point estimates of the primary endpoint, as well as the ability to observe rare adverse events or complications.

Assuming the primary endpoint of VT incidence is 10% for a specific type of device, with a sample size of 150, the precision of the point estimate is 4.8% (i.e. the 95% confidence interval is the point estimate plus/minus 4.8%).

Additionally, with a sample size of 150, the probability of observing at least one rare AE/complication with a 1% rate is 78% and the probability of observing at least one rare AE/complication with a 2% rate is 95%.

A sample size of 150 is proposed for each type of device (PowerPICC, PowerPICC SOLO, and PowerGroshong PICC) for a total of 450 participants in the study.

#### 1.3 Interim Analysis

An interim analysis, to assess study progress, will be targeted when 50% of the subjects have completed the study, or sooner, based on reporting requirements. As all analyses are only exploratory and no confirmatory tests are planned no alpha adjustment for the interim analysis is needed.

#### 1.4 Objectives

The primary safety objective is to assess the incidence of symptomatic venous thrombosis (VT) in patients with PowerPICC, PowerPICC SOLO, and PowerGroshong PICC devices (PICCs) used for both short- and long-term venous access.

The primary performance objective is to assess the rate of therapy completion in PICCs used for both short- and long-term therapy.



#### 2 Safety and Performance Variables

#### 2.1 Primary Safety Variable

The primary safety parameter for this study is the incidence of symptomatic VT defined as any new occurrence of symptomatic VT defined by thrombus presence confirmed by ultrasonography or other imaging.

#### 2.2 Primary Performance Variable

The primary performance parameter for this study is the percent of PICCs that remain in place through the required therapy time period (completion of therapy) (success/failure)

#### 2.3 Secondary Safety Variables

The following secondary safety parameters will be analyzed:

Incidence defined as any new occurrence of:

| Phlebitis |
|----------------------------------------|
| Extravasation |
| Local infection |
| Catheter-related bloodstream infection |
| Accidental dislodgement |
| Vessel laceration |

#### 2.4 Secondary Performance Variables

Vessel perforation

The following secondary performance parameters will be analyzed:

- Percent of patent catheters (number of functional catheters through therapy/total number of catheters)
- Percent of placement success in single insertion attempt (placement success defined as single insertion attempt, proper tip location, and patent catheter) (successful placement / total insertions)
- □ Usability: Ease of insertion based on a post-insertion survey

#### 2.5 Further Safety Variables

- Adverse events
- Device deficiencies



#### 3 Statistical Analysis Sets

#### 3.1 Enrolled Set

The enrolled set (ES) consists of all participants who sign the ICF.

#### 3.2 Safety Set

The safety set (SAF) consists of all participants who undergo placement of a study device.

#### 3.3 Evaluable Set

The evaluable set (EVS) consists of all participants who undergo successful placement of a study device and receive at least one treatment through it.

#### 3.4 Additional Subgroup Analysis

All analyses will be presented separately for the type of device (PowerPICC, PowerPICC SOLO, and PowerGroshong PICC).

#### 3.5 Assignment of Analysis Sets to Analysis

The evaluable set will be considered the primary analysis set for the primary performance endpoint. Disposition data will be analyzed on the enrolled set. Demographic data and safety analyses are presented using the safety set.



#### 4 Statistical Evaluation

The three types of devices (PowerPICC, PowerPICC SOLO, and PowerGroshong PICC) will be separately tabulated. Total columns will additionally be displayed for all three different types of devices combined.

No inferential assessments will be performed on any analyzed data.

A detailed description of the planned tables, listings and graphs is given in Appendix A (version 5.0).

#### 4.1 **Dispositions of Participants and Analysis Sets**

treatment with cervical collars or halo traction

history of phlebitis

history of venous thrombosis

#### Disposition of participants and analysis sets

The disposition of participants and analysis sets, participants per center, participants per country, inclusion and exclusion criteria, and the status at study termination will be shown on the enrolled set.

#### 4.2 **Demographics and Other Covariates**

#### Demographic data

Demographic data (age (at signing informed consent), gender, race, body height, body weight, body mass index (BMI)) will be tabulated

#### Medical history

| The pro | portion of | partici | pants with |
|---------|------------|---------|------------|
|---------|------------|---------|------------|

| e pr | oportion of participants with |
|---|---|
| | implantable devices |
| | past and/or current use of an artificial heart |
| | past and/or current anatomical abnormalities of the central venous system |
| | past and/or current use of an atrial fibrillation or other atrial arrhythmias that affects the p-wave |
| | known ABSENCE of a p-wave |
| | abnormalities of the arms |
| | abnormalities of the chest wall |
| | history of coagulopathy |
| | history of hypercoagulopathy |
| | current treatment with anticoagulants |
| | central venous access devices |
| | history of lymph node dissection/ lymphedema |
| | renal impairment |



- history of deep vein thrombosis
- □ history of catheter related bloodstream infection
- any other relevant medical history

will be tabulated.

Further details of medical history and details of other relevant medical history will be listed.

#### Baseline information

The primary and secondary diagnosis for current admission and the reason for PICC placement as well as the intended access duration will be tabulated.

Demographics and other covariates will be presented for the safety set.

#### 4.3 Catheter insertion, Maintenance and Removal

#### Catheter insertion

The location of procedure performance (bedside/ interventional radiology) will be tabulated.

The following information regarding catheter insertion will be tabulated:

- Was the catheter tip repositioned?
- What device was placed?
- What guidewire was used to facilitate insertion?
- Where was the catheter placed?
- Which vein was accessed for the procedure?
- Was an assessment of the vessel/catheter ratio done prior to insertion?
- □ How many insertion attempts were made?
- Was local anaestesia used?
- Was the catheter length trimmed?
- □ Was the insertion of the catheter done using tunneling?
- Was a Sherlock TLS used for placement?
- Was a Sherlock 3CG used for placement?
- □ What method was used to confirm catheter tip positioning?
- □ What stabilization method was used?
- What dressing type was used?
- □ Was the catheter inserted as per the instructions for use?
- □ Was a second implanted line vascular access device present (together with location and type of second device)?

Basic statistics for the duration between start and PICC is secured and the duration between start and tip position confirmation will be displayed. All catheter insertion data will be presented on the safety set.



#### Use and Maintenance

All information about participant location will be listed.

#### Removal

The proportion of participants with study PICC still in place, the reason for PICC removal, the proportion of participants with skin condition around the catheter site normal at removal and the specification of abnormal skin condition, and the use of the PICC line during the study period will be tabulated. Removal data will be presented for the evaluable set.

#### 4.4 Safety Analysis

All primary and secondary safety parameters will be analyzed using descriptive methods. For proportions exact two-sided 95% Clopper-Pearson confidence intervals will be calculated where appropriate. All safety analyses will be based on the safety set.

#### 4.4.1 Analysis of Primary Safety Variable

The primary safety endpoint for this study is the incidence of symptomatic VT defined as any new occurrence of symptomatic VT defined by thrombus presence confirmed by ultrasonography or other imaging.

The incidence rate of symptomatic VT will be calculated as the number of participants with symptomatic VT incidence (as ticked on the AE CRF page) divided by the total number of participants with non-missing data on symptomatic VT in the safety set and displayed using frequency tables. 95% confidence interval for the incidence rate will be additionally presented.

#### 4.4.2 Analysis of Secondary Safety Variables

#### **Complications**

For each complication listed as a secondary endpoint, the incidence will be calculated by dividing the number of participants experiencing the event by the total number of participants with non-missing data on the corresponding complication in the safety set and displayed using frequency tables. 95% confidence interval for the incidence will be additionally presented.

The following complications will be analyzed:

- □ Phlebitis (Preferred term (PT): "Catheter site phlebitis" / Lower level term (LLT): "Catheter site phlebitis")
- □ Extravasation (PT: "Catheter site extravasation" / LLT: "Catheter site extravasation")
- □ Local infection (as ticked on the adverse event (AE) case report form (CRF) page)
- Catheter-related bloodstream infection (as ticked on the AE CRF page)
- □ Accidental dislodgement (System organ class (SOC): "Product issues" / PT: "Device dislocation" / LLT: "Catheter dislodgment")
- Vessel laceration (as recorded on the catheter insertion CRF page)
- Vessel perforation (as recorded on the catheter insertion CRF page)

For local infections additionally the number of participants with local infections confirmed according to protocol (presence of pus at the exit site and/or culture confirmed site infection) by type of device and overall will be displayed in a footnote.



#### 4.4.3 Further Safety Variables

#### Adverse events (AEs)

AEs will be coded by using the Medical dictionary for regulatory activities version 23.0 (MedDRA).

AEs will be tabulated by SOC and PT (MedDRA). The number of entries, as well as the number and rate of affected participants will be reported for each type of device. Additionally, AEs will be presented by severity.

SAEs, non-serious AEs, and AEs which are related to device (adverse device effects [ADEs]), SADEs, AEs which are related to procedure, or related to accessories will be presented separately.

All AEs will be listed together with study day of AE (start date of AE – insertion date) as well as duration of AE for AEs with complete dates.

AEs are considered being related to device/procedure/accessories, if relationship is at least likely or relationship assessment is missing.

#### Device deficiencies

Details regarding device deficiencies will be listed.

#### 4.5 Performance Analysis

All primary and secondary performance parameters will be analyzed using descriptive methods. For proportions two-sided exact 95% Clopper-Pearson confidence intervals will be calculated where appropriate.

#### 4.5.1 Analysis of Primary Performance Variable

The primary performance parameter for this study is the percent of PICCs that remain in place through the required therapy time period (completion of therapy) (success/failure). A success will be defined as follows:

- subjects which still have the study peripherally inserted central line catheter in place
- subjects who did not have the study peripherally inserted central line catheter in place with the reason for peripherally inserted central line catheter removal:
  - "therapy completed / end of useful medical use (catheter stayed in place through the required therapy time)" or
  - "therapy changed or cancelled".

The percentage of PICCs that remain in place through the completion of therapy (success) will be calculated by dividing successful cases by the total number of devices with non-missing data on success/failure in the evaluable set and displayed using frequency tables. 95% confidence interval will be calculated.

#### 4.5.2 Analysis of Secondary Performance Variables

#### Percent of patent catheters

The percent of patent catheters will be calculated by dividing the number of catheters remaining functional through completion of therapy by the total number of catheters with non-missing data on patency in the evaluable set and displayed using frequency tables. 95% confidence intervals will be additionally calculated.



#### Percent of placement success in single insertion attempt

The percent of placement success in a single insertion attempt will be calculated by dividing the number of catheters that are placed in a single attempt with proper tip location, and catheter patency by the total number of insertions with non-missing data on placement success and number of attempts and displayed using frequency tables. 95% confidence intervals will be additionally calculated. Data will be presented on the safety set.

#### Usability: Ease of insertion - based on a post-insertion survey

The usability of guidewires/stylets will be analyzed based on a composite score of performance questions administered in a post-insertion survey.

The results of the insertion user questionnaire will be tabulated. For each question, the individual results will be tabulated. Additionally, for all scores, a numerical score will be applied (5 = very easy / strongly agree; 1 = very difficult / strongly disagree) and basic statistics will be additionally presented. Data will be presented on the safety set. Cases where the use of Sherlock TLS or 3CG is documented with "No" and no documentation is available in the ease of insertion data ("empty CRF documentation") for the respective question, will be displayed as "not applicable/not used" for the corresponding question.

#### 4.6 Other Analysis

#### Protocol deviation

Details regarding protocol deviations will be listed.

#### 4.7 Missing Values

No missing value imputation methods will be applied. During the data review meeting (DRM) all participants will be reviewed regarding their occurrence of missing data on safety and performance endpoints.

#### 4.8 Interim Analysis

All parameters captured on CRF pages belonging to data of participants needed for the interim analysis will be checked, as specified in the data validation plan and all queries will be resolved. The interim analysis will be performed at the time when 50% of the patients are enrolled. A cut-off date for the interim analysis will be fixed and all assessments done until the cut-off date will be entered in the eCRF and cleaned for the interim analysis. Only these data will be used for the interim analysis. Further unclean data entered in the eCRF will be cut and not used for the interim analysis.

As all analyses are only exploratory and no confirmatory tests are planned no alpha adjustment for the interim analysis is needed.

#### 4.9 Data Base Closure and Data Review

A data base closure will be performed prior to the final analysis. All parameters will be checked, as specified in the data validation plan, and all queries resolved before data base closure and final analysis.

A data snapshot will be done for the interim analysis.



A data review will be conducted prior to the interim and final analysis on all data to allocate the participants to the analysis sets. At least the following items will be discussed:

- □ Successful placement of a study device [listing 3.1]
- □ Receipt of at least one treatment through study device [listing 3.5]

These evaluations and assessments will be done together and in agreement with the Sponsor, however FGK will provide the Sponsor with the appropriate participant listings (as defined in appendix A). Data review can be done via a telephone conference or in writing.

The affiliation of participants to the analysis sets will be done prior to the analysis.

Data analysis will be done after data base closure and data review has been conducted and data review minutes have been signed by both the Sponsor and FGK.

#### 4.10 Miscellaneous

The description of the tables in Appendix A determines the general format of the tables. The real design will be determined by the technical possibilities within SAS and may not look identical to the provided example. However, all information as displayed will be included.

For qualitative variables frequency tables (absolute and relative values) will be presented. For frequency tables, all missing values (including user-defined missing values) will be displayed in one combined category "missing", but not included in the calculation of percentages. Percentages will be presented to one decimal place. Quantitative parameters will be described by declaring the mean value, standard deviation, minimum, first quartile, median, third quartile, and maximum. In general, minimum and maximum will be presented to the same level of precision as the raw data; means and medians, and quartiles will be presented to one further decimal place; standard deviations will be printed out to one additional place further. In basic statistics tables the overall number of missing values (including user-defined missing values as "not done", "unknown", "not applicable", "not documented") will be given.

The listings are always sorted by type of device, center, and participant. If a different sorting order should be used for some listings this will be remarked separately. The variables for the special listings are explicitly given in the description of listings. All listings will be presented for the safety set and an indicator if the patient is also in the evaluable set will be added to all listings, if not stated differently.

Enrolled participants without placement of device will be considered in tables and listings describing disposition of participants, analysis sets, and inclusion and exclusion criteria. Protocol deviations will be listed for enrolled patients.

The following title will be used for all generated tables, listings, and graphs for the interim/ final analysis:

Becton Dickinson Page # of #

Protocol: MDS-19PICCEU01 - <Interim/Final> Analysis



The numbering NNN of the tables/listings/graphs will be stated in the detailed description (Appendix A).

Following footnote will be used for all generated tables, listings, and graphs:

Program name: <Name of program> Date: <Actual date(DDMMMYYYY:hhmmss)>

All tables, listings, and graphs will be generated in A4 paper format.

The statistical evaluation will be performed using SAS version 9.4 or higher.

#### 5 Changes from Protocol

In the protocol the calculation of percentages for the safety and performance endpoints is described as dividing the numbers of participants with events by the total number of participants. This was corrected in the SAP to dividing by the number of participants with non-missing data for the respective endpoints only.



#### 6 Signatures

This SAP will be signed electronically in the eTMF.

#### Statistician:

Petra Wolf

Senior Statistician

FGK Clinical Research GmbH

Heimeranstr. 35

80339 München

Germany

#### Sponsor:

Gloria Viti

Clinical Project Manager

**Becton Dickinson and Company** 

Via Enrico Cialdini, 16

20161 Milan

Italy

#### Sponsor:

Rachel Gao

Senior Statistician

Becton Dickinson and Company

1 Becton Drive, Franklin Lakes,

New Jersey 07417

United States

# Statistical Analysis Plan Appendix A

List of generated summary tables, listings, and graphs

Version 5.0

Tables and listing needed for the interim analysis are marked with (\*)

#### **Table of Contents**

| TAE | BLE OF CONTENTS | 2 |
|---|---|---|
| 1 | DISPOSITION OF PARTICIPANTS | ı |
| 1.1 | Disposition of Participants / Analysis Sets | |
| | Table 1.1.1: Participants per Type of Device and Analysis Set | |
| | Table 1.1.2: Participants per Analysis Set and Center | |
| | Table 1.1.3: Participants per Analysis Set and Device | |
| | Table 1.1.4: Participants per Analysis Set and Country | |
| | Table 1.1.5: Inclusion and Exclusion Criteria | |
| | Listing 1.1.1: Disposition of Participants and Analysis Sets | |
| 1.2 | Discontinuation | |
| | Table 1.2.1: Status at End of Study (*) | |
| | Listing 1.2.1: Study Termination | |
| • | | |
| 2 | DEMOGRAPHIC DATA AND OTHER COVARIATES | |
| | Table 2.1: Participant Demographics – Frequencies Table 3.2: Participant Demographics – Regio Statistics | |
| | <ul> <li>Table 2.2: Participant Demographics – Basic Statistics</li> <li>Listing 2.1: Participant Demographics</li> </ul> | |
| | Listing 2.2: Medical History Listing 2.3: Other Medical History | |
| | Table 2.4: Baseline Information | |
| | Listing 2.4: Baseline Information | |
| 3 | CATHETER INSERTION, MAINTENANCE AND REMOVAL | |
| | Table 3.1: Catheter Insertion: Procedure Details | |
| | Table 3.2: Catheter Insertion: Duration | |
| | Listing 3.1: Catheter Insertion: Procedure Details | |
| | Table 3.3: Catheter Insertion: Device | |
| | Listing 3.2: Catheter Insertion: Device | |
| | Listing 3.3: Catheter Insertion: Additional Kits | |
| | Table 3.4: Catheter Insertion: Insertion | |
| | Listing 3.4: Catheter Insertion: Insertion (*) | 52 |

| | Listing 3.5: Participant Location | 53 |
|---|---|---|
| | Table 3.5: Removal | 54 |
| | Listing 3.6: Removal (*) | |
| | Listing 3.7: Removal: Complications and Performance (*) | 58 |
| 4 | SAFETY | 59 |
| 4.1 | Primary Safety Variable | 59 |
| | Table 4.1.1: Incidence of Symptomatic Venous Thrombosis (*) | 60 |
| 4.2 | · · | |
| 4. | 4.2.1 Complications | 61 |
| | Table 4.2.1.1: Complications (*) | 62 |
| 4.3 | Further Safety Variables | 69 |
| 4. | 4.3.1 Adverse Events | 69 |
| | Table 4.3.1.1: Number of Participants with (S)AEs, (S)ADEs, and Related AEs | 70 |
| | Table 4.3.1.2: AEs by System Organ Class | 71 |
| | Table 4.3.1.3: AEs by System Organ Class and Severity | 72 |
| | Table 4.3.1.4: Serious AEs by System Organ Class | |
| | Table 4.3.1.5: Non-serious AEs by System Organ Class | 74 |
| | Table 4.3.1.6: Adverse Device Effects by System Organ Class | 75 |
| | Table 4.3.1.7: Serious Adverse Device Effects by System Organ Class | |
| | Table 4.3.1.8: AEs Related to Procedure by System Organ Class | 77 |
| | Table 4.3.1.9: AEs Related to Accessories by System Organ Class | 78 |
| | Listing 4.3.1.1: Adverse Events (*) | |
| | Listing 4.3.1.2: Serious Adverse Events - AE Form | |
| | Listing 4.3.1.3: Serious Adverse Events - SAE Form | |
| 4. | 4.3.2 Device Deficiencies | |
| | Listing 4.3.2.1: Device Deficiencies | 83 |
| 5 | PERFORMANCE ANALYSIS | 84 |
| 5.1 | Analysis of Primary Performance Variable | 84 |
| | Table 5.1.1: PICCs that remain in place through completion of therapy (*) | 85 |
| 5.2 | | |
| | Table 5.2.1: Patent Catheters (*) | 87 |

## **Interim and Final Analysis**

## Appendix A


| | Table 5.2.2: Placement Success in Single Insertion Attempt (*) | 88 |
|---|---|---|
| | Table 5.2.3: Usability: Ease of Insertion – Guidewire (*) | |
| | Table 5.2.4: Usability: Ease of Insertion – Guidewire – Basic Statistics (*) | |
| | Table 5.2.5: Usability: Ease of Insertion – Stylet (*) | 94 |
| | Table 5.2.6: Usability: Ease of Insertion – Stylet – Basic Statistics (*) | |
| | Listing 5.2.1: Usability: Ease of Insertion – Guidewire (*) | |
| | Listing 5.2.2: Usability: Ease of Insertion – Stylet (*) | |
| 6 | PROTOCOL DEVIATIONS | |
| • | Listing 6.1: Protocol Deviations (eCRF) | |

Statistical Analysis Plan MDS-19PICCEU01

- 1 Disposition of Participants
- 1.1 Disposition of Participants / Analysis Sets

 Table 1.1.1: Participants per Type of Device and Analysis Set Enrolled Set

Statistical Analysis Plan MDS-19PICCEU01

| | Type of Device | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| | PowerPICC<br>(N=XXX) | | PowerPICC SOLO (N=XXX) | | PowerGroshong PICC (N=XXX) | | Device Not Assigned (N=3) | Total<br>(N=XXX) | |
| Enrolled Set (ES) | N | % | N | % | N | % | | N | % |
| no | | | | | | | | | |
| yes | | | | | | | | | |
| Overall (non-missing) | | | | | | | | | |

| | Type of Device | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| | PowerPICC<br>(N=XXX) | | PowerPICC SOLO (N=XXX) | | PowerGroshong PICC (N=XXX) | | Device Not Assigned (N=3) | Total<br>(N=XXX) | |
| Safety Set (SAF) | N | % | N | % | N | % | | N | % |
| no | | | | | | | | | |
| yes | | | | | | | | | |
| Overall (non-missing) | | | | | | | | | |

| | | Type of Device | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| | PowerPICC<br>(N=XXX) | | PowerPICC SOLO (N=XXX) | | PowerGroshong PICC (N=XXX) | | Device Not Assigned (N=3) | Total<br>(N=XXX) | |
| Evaluable Set (EVS) | N | % | N | % | N | % | | N | % |
| no | | | | | | | | | |
| yes | | | | | | | | | |
| Overall (non-missing) | | | | | | | | | |

Footnote 1: For the subsequent tables, listings, and graphs, only the short labels for the statistical analysis sets (given in brackets) are used.

• Table 1.1.2: Participants per Analysis Set and Center

#### **Enrolled Set**

| | Analysis Set | | | | | |
|---|---|---|---|---|---|---|
| | | ed Set<br>(XX) | | ible Set<br>XXX) | Safety Set<br>(N=XXX) | |
| Center | N | % | N | % | N | % |
| 1 | | | | | | |
| 2 | | | | | | |
| 3 | | | | | | |
| 4 | | | | | | |
| Overall (non-missing) | | | | | | |

• Table 1.1.3: Participants per Analysis Set and Device

#### **Enrolled Set**

| | | | Analys | sis Set | | |
|---|---|---|---|---|---|---|
| | Enrolled Set<br>(N=XXX) | | | Evaluable Set<br>(N=XXX) | | y Set<br>(XX) |
| Device | N | % | N | % | N | % |
| missing | | | | | | |
| PowerPICC | | | | | | |
| PowerPICC SOLO | | | | | | |
| PowerGroshong PICC | | | | | | |
| Device Not Assigned | | | | | | |
| Overall (non-missing) | | | | | | |

• Table 1.1.4: Participants per Analysis Set and Country

#### **Enrolled Set**

| | Analysis Set | | | | | |
|---|---|---|---|---|---|---|
| | | ed Set<br>XXX) | Evaluable Set<br>(N=XXX) | | Safety Set<br>(N=XXX) | |
| Country | N | % | N | % | N | % |
| Overall (non-missing) | | | | | | |

#### • Table 1.1.5: Inclusion and Exclusion Criteria

#### **Enrolled Set**

| | | | | | Type of | Device | | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| | Powe | rPICC | PowerPIC | CC SOLO | PowerGros | hong PICC | Device No | t Assigned | То | tal |
| | (N=) | (N=xxx) | | xxx) | (N=xxx) | | (N=3) | | (N=xxx) | |
| All inclusion criteria met | N | % | N | % | N | % | | | N | % |
| no | | | | | | | | | | |
| yes | | | | | | | | | | |
| Overall (non-missing) | | | | | | | | | | |

| | | | | | Type of | Device | | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| | Powe | rPICC | PowerPIC | CC SOLO | PowerGros | hong PICC | Device Not Assigned | | Total | |
| | (N=) | (N=xxx) | | N=xxx) (N=xxx) | | (N=3) | | (N=xxx) | | |
| None of the exclusion criteria met | N | % | N | % | N | % | | | N | % |
| no | | | | | | | | | | |
| yes | | | | | | | | | | |
| Overall (non-missing) | | | | | | | | | | |

| | | | | | Type of | Device | | | |
|---|---|---|---|---|---|---|---|---|---|
| | Powe | rPICC | PowerPIC | CC SOLO | PowerGros | hong PICC | Device Not Assigned | Total | |
| | (N=) | (N=xxx) | | xxx) | (N=xxx) | | (N=3) | (N=xxx) | |
| All inclusion criteria<br>and none of the<br>exclusion criteria met | N | % | N | % | N | % | | N | % |
| no | | | | | | | | | |
| yes | | | | | | | | | |
| Overall (non-missing) | | | | | | | | | |

• Listing 1.1.1: Disposition of Participants and Analysis Sets

**Enrolled Set** 

**Variables**: Type of device, Center, Country, Participant, ICF version date, Date/Time ICF signed, All IC and EC met (yes/no), Violated IC^, Violated EC^, Agreed to use the study data for further research, Subject status, EVS (yes/no), SAF (yes/no)

Footnote 1: ^ Numbers (eCRF) of violated IC or EC.

Note: Type of device will be displayed as "by-variable" within a subtitle.

1.2 Discontinuation

• Table 1.2.1: Status at End of Study (\*)

Safety Set

| | Type of Device | | | | | | | |
|---|---|---|---|---|---|---|---|---|
| | | rPICC<br>xxx) | | CC SOLO | PowerGroshong PICC<br>(N=xxx) | | Total<br>(N=xxx) | |
| Completion status (CRF) | N | % | N | % | N | % | N | % |
| missing | | | | | | | | |
| completed (removal and/or 180 days) | | | | | | | | |
| withdrawal | | | | | | | | |
| Overall (non-missing) | | | | | | | | |

| | | | | Type of | Device | | | |
|---|---|---|---|---|---|---|---|---|
| | | PowerPICC<br>(N=xxx) | | CC SOLO | PowerGroshong PICC<br>(N=xxx) | | | otal<br>xxx) |
| Reason for withdrawal | N | % | N | % | N | % | N | % |
| missing | | | | | | | | |
| withdrawal of consent | | | | | | | | |
| lost to follow up | | | | | | | | |
| death | | | | | | | | |
| AE | | | | | | | | |
| device deficiency | | | | | | | | |
| other | | | | | | | | |
| Overall (non-missing) | | | | | | | | |

Note 1: Reason for withdrawal only displayed for patients with study withdrawal.

| | | | | Type of | Device | | | | |
|---|---|---|---|---|---|---|---|---|---|
| | Power<br>(N=x | | | | | | PowerGroshong PICC<br>(N=xxx) | | Total<br>(N=xxx) |
| Completion status | N | % | N | % | N | % | N | % | |
| missing | | | | | | | | | |
| completed (removal and/or 180 days) | | | | | | | | | |
| death | | | | | | | | | |
| lost to follow up | | | | | | | | | |
| withdrawal | | | | | | | | | |
| Overall (non-missing) | | | | | | | | | |

• Listing 1.2.1: Study Termination

Safety Set

Variables: Type of device, Participant, Date of study completion, Completion status, Reason for withdrawal, Specification of other reason,

Date of death, EVS (yes/no), SAF (yes/no)

Note: Type of devices will be displayed as "by-variable" within a subtitle.

2 Demographic Data and Other Covariates

• Table 2.1: Participant Demographics – Frequencies

Safety Set

| | Type of Device | | | | | | | |
|---|---|---|---|---|---|---|---|---|
| | Powe | rPICC | PowerPICC SOLO PowerGroshong PICC | | Total | | | |
| | (N= | xxx) | (N= | xxx) | (N=xxx) | | (N=xxx) | |
| Gender | N % | | N | % | N | % | N | % |
| missing | | | | | | | | |
| male | | | | | | | | |
| female | | | | | | | | |
| Overall (non-missing) | | | | | | | | |

| | | | | Type of | Device | | | |
|---|---|---|---|---|---|---|---|---|
| | PowerPICC | | PowerPlo | CC SOLO | PowerGroshong PICC | | Total | |
| | (N=x | (XX) | (N= | xxx) | (N=) | xxx) | (N= | xxx) |
| Race | N | % | N | % | N | % | N | % |
| missing | | | | | | | | |
| White | | | | | | | | |
| Asian | | | | | | | | |
| Black or African American | | | | | | | | |
| other | | | | | | | | |
| unknown | | | | | | | | |
| Overall (non-missing) | | | | | | | | |

FGK

 Table 2.2: Participant Demographics – Basic Statistics Safety Set

| | | | Type of Device | | Total |
|---|---|---|---|---|---|
| | | PowerPICC<br>(N=xxx) | PowerPICC SOLO (N=xxx) | PowerGroshong PICC (N=xxx) | (N=xxx) |
| | N | | | | |
| | missing | | | | |
| | mean | | | | |
| | SD | | | | |
| Age [years]^ | minimum | | | | |
| | 1st quartile | | | | |
| | median | | | | |
| | 3rd quartile | | | | |
| | maximum | | | | |

#### **Footnote 1:** ^ Age at signing informed consent.

| | | | Type of Device | Total |
|---|---|---|---|---|
| | | PowerPICC PowerPICC SOLO PowerGroshong PICC (N=xxx) (N=xxx) | | |
| | N | | | |
| | missing | | | |
| | mean | | | |
| | SD | | | |
| Body height [cm] | minimum | | | |
| | 1st quartile | | | |
| | median | | | |
| | 3rd quartile | | | |
| | maximum | _ | | |

| | 1 | - |
|------------------|--------------|---|
| Body weight [kg] | N | |
| | missing | |
| | mean | |
| | SD | |
| | minimum | |
| | 1st quartile | |
| | median | |
| | 3rd quartile | |
| | maximum | |
| BMI [kg/m²] | N | |
| | missing | |
| | mean | |
| | SD | |
| | minimum | |
| | 1st quartile | |
| | median | |
| | 3rd quartile | |
| | maximum | |

• Listing 2.1: Participant Demographics

Safety Set

**Variables:** Type of device, Participant, Age [years]^, Gender, Race (including specification of other race), Body height [cm], Body weight [kg], BMI [kg/m2], Evaluable Set (yes/no)

**Footnote 1:** ^ Age at signing informed consent.

# • Table 2.3: Medical History

### Safety Set

| | | | | Type of | Device | | | |
|---|---|---|---|---|---|---|---|---|
| | Powe | rPICC | PowerPl | CC SOLO | PowerGros | shong PICC 1 | | otal |
| | (N= | xxx) | (N= | xxx) | (N= | xxx) | (N=xxx) | |
| Implantable devices | N | N % | | % | N | % | N | % |
| missing | | | | | | | | |
| no | | | | | | | | |
| yes | | | | | | | | |
| Overall (non-missing) | | | | | | | | |

| | | | | Type of | Device | | | |
|---|---|---|---|---|---|---|---|---|
| | PowerPICC | | PowerPICC SOLO | | PowerGros | hong PICC | Total<br>(N=xxx) | |
| | (N= | (N=xxx) | | xxx) | (N=xxx) | | | |
| Past and/or current use of an artificial heart | N | % | N | % | N | % | N | % |
| missing | | | | | | | | |
| no | | | | | | | | |
| yes | | | | | | | | |
| Overall (non-missing) | · | | | | | | | |

| | | | | Type of | Device | | | |
|---|---|---|---|---|---|---|---|---|
| | Powe | rPICC | PowerPi | CC SOLO | PowerGros | werGroshong PICC | | otal |
| | (N=) | xxx) | (N=: | xxx) | (N=xxx) (N=xxx) | | xxx) | |
| Past and/or current anatomical abnormalities of the central venous system | N | % | N | % | N | % | N | % |
| missing | | | | | | | | |
| no | | | | | | | | |
| yes | | | | | | | | |
| Overall (non-missing) | | | | | | | | |

| | | | | Type of | Device | | | |
|---|---|---|---|---|---|---|---|---|
| | Powe | rPICC | PowerPl | CC SOLO | PowerGroshong PICC | | To | tal |
| | (N= | xxx) | (N= | xxx) | (N=xxx) (N=xxx) | | | xxx) |
| Past and/or current use of an atrial fibrillation or other atrial arrhythmias that affects the p-wave | N | % | N | % | N | % | N | % |
| missing | | | | | | | | |
| no | | | | | | | | |
| yes | | | | | | | | |
| Overall (non-missing) | | | | | | | | |

| | | | | Type of | Device | | | |
|---|---|---|---|---|---|---|---|---|
| | Powe | rPICC | PowerPl | CC SOLO | PowerGros | verGroshong PICC T | | otal |
| | (N= | xxx) | (N= | xxx) | (N= | xxx) | (N=xxx) | |
| Known absence of a p-wave | N % | | N | % | N % N | | N | % |
| missing | | | | | | | | |
| no | | | | | | | | |
| yes | | | | | | | | |
| Overall (non-missing) | | | | | | | | |

| | | | | Type of | Device | | |
|---|---|---|---|---|---|---|---|
| | | rPICC | | | otal | | |
| | (N= | xxx) | (N= | xxx) | (N=xxx) | (N= | vtal<br>xxx)<br>% |
| Abnormalities of the arms | N % | | N | % | N % | N | % |
| missing | | | | | | | |
| no | | | | | | | |
| yes | | | | | | | |
| Overall (non-missing) | | | | | | | |

| | | | Type of Device | | | | |
|---|---|---|---|---|---|---|---|
| | Powe | rPICC | PowerPi | CC SOLO | | То | otal |
| | (N= | xxx) | (N= | xxx) | | (N=xxx) | |
| Abnormalities of the chest wall | N % | | N | % | N % N | % | |
| missing | | | | | | | |
| no | | | | | | | |
| yes | | | | | | | |
| Overall (non-missing) | | | | | | | |

| | | | | Type of | Device | | |
|---|---|---|---|---|---|---|---|
| | Powe | rPICC | PowerPl | CC SOLO | PowerGros | shong PICC | Total<br>(N=xxx) |
| | (N= | xxx) | (N= | xxx) | (N= | xxx) | |
| History of coagulopathy | N % | | N | % | N % N | | % |
| missing | | | | | | | |
| no | | | | | | | |
| yes | | | | | | | |
| Overall (non-missing) | | | | | | | |

| | | | | Type of | Device | | | |
|---|---|---|---|---|---|---|---|---|
| | Powe | rPICC | PowerPi | CC SOLO | PowerGroshong PICC | | То | otal |
| | (N= | xxx) | (N= | xxx) | (N= | xxx) | (N= | xxx) |
| History of hypercoagulopathy | N % | | N | % | N % | | N | % |
| missing | | | | | | | | |
| no | | | | | | | | |
| yes | | | | | | | | |
| Overall (non-missing) | | | | | | | | |

| | | | | Type of | Device | | | Total<br>(N=xxx)<br>N % |
|---|---|---|---|---|---|---|---|---|
| | | rPICC<br>xxx) | | CC SOLO | | shong PICC | | |
| Current treatment with anticoagulants | N % | | N | % | , , | | , | |
| missing | | | | | | | | |
| no | | | | | | | | |
| yes | | | | | | | | |
| Overall (non-missing) | | | | | | | | |

| | | Type of Device PowerPICC PowerPICC SOLO PowerGroshong PICC Total (N=xxx) (N=xxxx) (N=xxxx) (N=xxxx) (N=xxxx) (N=xxxxx) (N=xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx | | | | | | |
|---|---|---|---|---|---|---|---|---|
| | (N= | xxx) | (N= | xxx) | (N= | xxx) | (N= | (N=xxx) |
| Central venous access devices | N % | | N | % | N % | | N | % |
| missing | | | | | | | | |
| no | | | | | | | | |
| yes | | | | | | | | |
| Overall (non-missing) | | | | | | | | |

| | | | | Type of Device PowerPICC SOLO PowerGroshong PICC Total (N=xxx) (N=xxx) (N=xxx) N % N % | | | | |
|---|---|---|---|---|---|---|---|---|
| | Powe | rPICC | PowerPl | PowerPICC SOLO PowerGroshong PICC | | То | otal | |
| | (N= | xxx) | (N= | xxx) | (N= | xxx) | (N= | xxx) |
| History of lymph<br>node dissection/<br>lymphedema | N | % | N | % | N | % | N | % |
| missing | | | | | | | | |
| no | | | | | | | | |
| yes | | | | | | | | |
| Overall (non-missing) | | | | | | | | |

| | Type of Device | | | | | | | |
|---|---|---|---|---|---|---|---|---|
| | PowerPICC<br>(N=xxx) | | PowerPl | CC SOLO | PowerGros | hong PICC | To | otal |
| | | | (N=xxx) | | (N=xxx) | | (N=xxx) | |
| Renal impairment | N | N % | | % | N | % | N | % |
| missing | | | | | | | | |
| no | | | | | | | | |
| yes | | | | | | | | |
| Overall (non-missing) | | | | | | | | |

| | | | Type of | Device | | | |
|---|---|---|---|---|---|---|---|
| | PowerPICC (N=xxx) N % | PowerPl | CC SOLO | PowerGros | hong PICC | Total | |
| | | (N=xxx) | | (N=xxx) | | (N=xxx) | |
| Treated with cervical collars or halo traction | | N | % | N | % | N | % |
| missing | | | | | | | |
| no | | | | | | | |
| yes | | | | | | | |
| Overall (non-missing) | | | | | | | |

| | Type of Device | | | | | |
|---|---|---|---|---|---|---|
| | PowerPICC<br>(N=xxx) | PowerPICC SOLO (N=xxx) | PowerGroshong PICC (N=xxx) | Total<br>(N=xxx) | | |
| | | | | | History of phlebitis | N % |
| missing | | | | | | |
| no | | | | | | |
| yes | | | | | | |
| Overall (non-missing) | | | | | | |

| | Type of Device | | | | | |
|---|---|---|---|---|---|---|
| | PowerPICC (N=xxx) N % | PowerPl | CC SOLO | PowerGros | shong PICC | Total |
| | | (N=xxx) | | (N=xxx) | | (N=xxx) |
| History of venous thrombosis | | N % | | N % | | N % |
| missing | | | | | | |
| no | | | | | | |
| yes | | | | | | |
| Overall (non-missing) | | | | | | |

| | | | | Type of | Device | | | |
|---|---|---|---|---|---|---|---|---|
| | PowerPICC<br>(N=xxx) | | PowerPl | CC SOLO | PowerGros | hong PICC | Тс | otal |
| | | | (N=xxx) | | (N=xxx) | | (N=xxx) | |
| History of deep vein thrombosis | N | N % | | % | N | % | N | % |
| missing | | | | | | | | |
| no | | | | | | | | |
| yes | | | | | | | | |
| Overall (non-missing) | | | | | | | | |

| | | | Type of | Device | | | |
|---|---|---|---|---|---|---|---|
| | PowerPICC (N=xxx) N % | PowerPi | CC SOLO | PowerGroshong PICC | | To | otal |
| | | (N=xxx) | | (N=xxx) | | (N=xxx) | |
| History of catheter related bloodstream infection | | N | % | N | % | N | % |
| missing | | | | | | | |
| no | | | | | | | |
| yes | | | | | | | |
| Overall (non-missing) | | | | | | | |

| | Type of Device | | | | | | |
|---|---|---|---|---|---|---|---|
| | PowerPICC<br>(N=xxx) | PowerPl | CC SOLO | PowerGros | hong PICC | To | otal |
| | | (N=xxx) | | (N=xxx) | | (N=xxx) | |
| Other relevant<br>Medical History | N % | N | % | N | % | N | % |
| missing | | | | | | | |
| no | | | | | | | |
| yes | | | | | | | |
| Overall (non-missing) | | | | | | | |

• Listing 2.2: Medical History

Safety Set

Variables: Type of device, Participant + all variables on medical history-form, Evaluable Set (yes/no)

• Listing 2.3: Other Medical History

Safety Set

FGK

Variables: Type of device, Participant, Sequence No., Term/Description, Start date, End date, Status (ongoing), Evaluable Set (yes/no)

Footnote 1: Only participants with at least one entry in 'Other Medical History' form are displayed.

## • Table 2.4: Baseline Information

Safety Set

| | | | | Type of | Device | | | |
|---|---|---|---|---|---|---|---|---|
| | Power | PowerPICC | | CC SOLO | PowerGroshong PICC | | Total | |
| | (N=xxx) | | (N=xxx) | | (N=xxx) | | (N=xxx) | |
| | N | % | N | % | N | % | N | % |
| Primary diagnosis for current admission | | | | | | | | |
| missing | | | | | | | | |
| cardiac | | | | | | | | |
| orthopedic | | | | | | | | |
| Overall (non-missing) | | | | | | | | |

| | | | | Type of | Device | | | |
|---|---|---|---|---|---|---|---|---|
| | Powe | erPICC | PowerPICC SOLO | | PowerGroshong PICC | | To | otal |
| | (N= | (N=xxx) | | (N=xxx) | | (N=xxx) | | xxx) |
| | N | % | N | % | N | % | N | % |
| Secondary<br>diagnosis for<br>current admission | | | | | | | | |
| missing | | | | | | | | |
| cardiac | | | | | | | | |
| orthopedic | | | | | | | | |
| Overall (non-missing) | | | | | | | | |

| | | | | | | Type of | Device | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | PowerPICC | | PowerPICC SOLO | | | PowerGroshong PICC | | | Total | | |
| | (N=xxx) | | (N=xxx) | | (N=xxx) | | | | (N=xxx) | | | |
| | Number of<br>Reasons | Reasons Part. with Reason | | | Number of<br>Part. with<br>Reason | Part. with<br>Reason | Number of<br>Reasons | Number of<br>Part. with<br>Reason | Part. with<br>Reason | Number of<br>Reasons | Number of<br>Part. with<br>Reason | Part. with<br>Reason |
| | (N#) | (N) | (%) | (N#) | (N) | (%) | (N#) | (N) | (%) | (N#) | (N) | (%) |
| Reason for PICC placement | | | | | | | | | | | | |
| limited peripheral access | | | | | | | | | | | | |
| IV therapy/pain management | | | | | | | | | | | | |
| Total | | | | | | | | | | | | |

| | | | | Type of | Device | | | |
|---|---|---|---|---|---|---|---|---|
| | Powe | PowerPICC<br>(N=xxx) | | CC SOLO | PowerGroshong PICC | | Total | |
| | (N= | | | (N=xxx) | | (N=xxx) | | xxx) |
| | N | % | N | % | N | % | N | % |
| Intended access duration | | | | | | | | |
| missing | | | | | | | | |
| short-term (<30 days) | | | | | | | | |
| long-term (>= 30 days) | | | | | | | | |
| Overall (non-missing) | | | | | | | | |

• Listing 2.4: Baseline Information

Safety Set

FGK

**Variables:** Type of device, Participant, Primary diagnosis for current admission / Specification of other, Secondary diagnosis for current admission / Specification of other, Reason for PICC placement / Specification of other reason, Intended access duration, Evaluable Set (yes/no)


3 Catheter Insertion, Maintenance and Removal

• Table 3.1: Catheter Insertion: Procedure Details

Safety Set

| | | | | Type of | Device | | | |
|---|---|---|---|---|---|---|---|---|
| | Power | PowerPICC<br>(N=xxx) | | PowerPICC SOLO (N=xxx) | | PowerGroshong PICC (N=xxx) | | otal |
| | (N=) | | | | | | | xxx) |
| | N | % | N | % | N | % | N | % |
| Location of procedure performance | | | | | | | | |
| missing | | | | | | | | |
| bedside | | | | | | | | |
| interventional radiology | | | | | | | | |
| other | | | | | | | | |
| Overall (non-missing) | | | | | | | | |

| | | | | Type of | Device | | | |
|---|---|---|---|---|---|---|---|---|
| | Powe | rPICC | PowerPl | PowerPICC SOLO | | hong PICC | Total | |
| | N % | | (N=xxx) | | (N=xxx) | | (N=xxx) | |
| | | | N | % | N | % | N | % |
| Catheter tip repositioning | | | | | | | | |
| missing | | | | | | | | |
| no | | | | | | | | |
| yes | | | | | | | | |
| Overall (non-missing) | | | | | | | | |

| | | | | Type of | Device | | | |
|---|---|---|---|---|---|---|---|---|
| | | PowerPICC<br>(N=xxx) | | CC SOLO | PowerGroshong PICC<br>(N=xxx) | | Total<br>(N=xxx) | |
| - | N | % | N | % | N (.t ) | % | N | % |
| Device placement successful | | | | | | | | |
| missing | | | | | | | | |
| no | | | | | | | | |
| yes | | | | | | | | |
| Overall (non-missing) | | | | | | | | |

• Table 3.2: Catheter Insertion: Duration

Safety Set

| | | | Type of Device | | Total |
|---|---|---|---|---|---|
| | | PowerPICC<br>(N=xxx) | PowerPICC SOLO (N=xxx) | PowerGroshong PICC (N=xxx) | Total<br>(N=xxx) |
| | N | | | | |
| | missing | | | | |
| Duration | mean | | | | |
| between | SD | | | | |
| start and<br>PICC is | minimum | | | | |
| secured | 1st quartile | | | | |
| [min] | median | | | | |
| | 3rd quartile | | | | |
| | maximum | | | | |

| | | | Type of Device | | Total |
|---|---|---|---|---|---|
| | | PowerPICC<br>(N=xxx) | PowerPICC SOLO (N=xxx) | PowerGroshong PICC (N=xxx) | Total<br>(N=xxx) |
| | N | | | | |
| | missing | | | | |
| Duration | mean | | | | |
| between | SD | | | | |
| start and tip position | minimum | | | | |
| confirmation | 1st quartile | | | | |
| [min] | median | | | | |
| | 3rd quartile | | | | |
| | maximum | | | | |


• Listing 3.1: Catheter Insertion: Procedure Details

Safety Set

**Variables:** Type of device, Participant, Where was the procedure performed / Specification, Insertion date, Procedure start time/stop time, Time of tip location confirmation, Duration between start and PICC is secured [min], Duration between start and tip position confirmation [min], Catheter tip repositioned, Device placement successful, Evaluable Set (yes/no)

• Table 3.3: Catheter Insertion: Device

Safety Set

| Device | Type of Device | | | | | | | |
|---|---|---|---|---|---|---|---|---|
| | PowerPICC<br>(N=xxx) | | PowerPICC SOLO (N=xxx) | | PowerGroshong PICC (N=xxx) | | Total<br>(N=xxx) | |
| | N | % | N | % | N | % | N | % |
| missing | | | | | | | | |
| PowerGroshong PICC-<br>Single - 5F- 40 cm | | | | | | | | |
| PowerGroshong PICC-<br>Single - 5F- 45 cm | | | | | | | | |
| Overall (non-missing) | | | | | | | | |

| | | | | Type of | Device | | | |
|---|---|---|---|---|---|---|---|---|
| | PowerPICC | | PowerPIC | CC SOLO | PowerGroshong PICC | | To | otal |
| (N=xxx) | | (N=xxx) | | (N=xxx) | | (N= | xxx) | |
| Guidewire | N % | | N | % | N | % | N | % |
| missing | | | | | | | | |
| BD nitinol 70 cm | | | | | | | | |
| BD nitinol 135 cm | | | | | | | | |
| Overall (non-missing) | | | | | | | | |

| | | | Type of | Device | | | |
|---|---|---|---|---|---|---|---|
| | PowerPICC (N=xxx) N % | PowerPICC SOLO (N=xxx) | | PowerGroshong PICC (N=xxx) | | Total<br>(N=xxx) | |
| Placement of catheter | | N | % | N | % | N | % |
| missing | | | | | | | |
| right arm | | | | | | | |
| left arm | | | | | | | |
| other | | | | | | | |
| Overall (non-missing) | | | | | | | |

| | | | | Type of | f Device | | | |
|---|---|---|---|---|---|---|---|---|
| | PowerPICC | | PowerPICC SOLO | | PowerGroshong PICC | | To | otal |
| (N=xxx) | | (N=xxx) | | (N=xxx) | | (N=xxx) | | |
| Vein | N % | | N | % | N | % | N | % |
| missing | | | | | | | | |
| basilic | | | | | | | | |
| cephalic | | | | | | | | |
| Overall (non-missing) | | | | | | | | |

| | | | Type of | Device | | | |
|---|---|---|---|---|---|---|---|
| | e prior to N % N % | PowerPICC SOLO | | PowerGroshong PICC | | Total | |
| | | (N=xxx) | | (N=xxx) | | | |
| Vessel/catheter ratio done prior to insertion | | N | % | N | % | N | % |
| missing | | | | | | | |
| no | | | | | | | |
| yes | | | | | | | |
| Overall (non-missing) | | | | | | | |

| | | | Type of | Device | | | |
|---|---|---|---|---|---|---|---|
| | N % | PowerPICC SOLO (N=xxx) | | PowerGroshong PICC<br>(N=xxx) | | Total<br>(N=xxx) | |
| Number of insertion attempts | | N | % | N | % | N | % |
| missing | | | | | | | |
| 1 | | | | | | | |
| 2 | | | | | | | |
| Overall (non-missing) | | | | | | | |

| | Type of Device | | | | |
|---|---|---|---|---|---|
| | PowerPICC (N=xxx) N % | PowerPl | CC SOLO | PowerGroshong PICC | Total |
| | | (N=xxx) | | (N=xxx) | (N=xxx) |
| Local anaesthesia used | | N % | | N % | N % |
| missing | | | | | |
| no | | | | | |
| yes | | | | | |
| Overall (non-missing) | | | | | |


• Listing 3.2: Catheter Insertion: Device

Safety Set

FGK

Variables: Type of device, Participant, What device was placed, What guidewire was used / Specification, Kit / tray catalog number, Kit / tray lot number, Kit / tray expiration date, More than 1 kit used, Where was catheter placed / Specification, Which vein was accessed / Specification, Assessment of the vessel/catheter ratio done, Vessel diameter, Vessel to catheter ratio, No. of insertion attempts, Local anaesthesia used, Evaluable Set (yes/no)

• Listing 3.3: Catheter Insertion: Additional Kits

Safety Set

**Variables:** Type of device, Participant, Sequence No., Kit / tray catalog number, Kit / tray lot number, Kit / tray expiration date, Implanted catheter from this kit, Guidewire used from this kit, Evaluable Set (yes/no)

• Table 3.4: Catheter Insertion: Insertion

Safety Set

| | Type of Device | | | | | | | |
|---|---|---|---|---|---|---|---|---|
| | PowerPICC<br>(N=xxx) | | PowerPICC SOLO (N=xxx) | | PowerGroshong PICC (N=xxx) | | Total<br>(N=xxx) | |
| Catheter length trimmed | N | N % | | % | N | % | N | % |
| missing | | | | | | | | |
| no | | | | | | | | |
| yes | | | | | | | | |
| Overall (non-missing) | | | | | | | | |

| | | | | Type of | Device | | | |
|---|---|---|---|---|---|---|---|---|
| | Powe | rPICC | PowerPICC SOLO | | PowerGroshong PICC | | Total | |
| | (N= | xxx) | (N= | xxx) | (N=xxx) | | (N= | xxx) |
| Tunneling used | N | % | N % N % | | N | % | | |
| missing | | | | | | | | |
| no | | | | | | | | |
| yes | | | | | | | | |
| Overall (non-missing) | | | | | | | | |

| | | Type of Device erPICC PowerPICC SOLO PowerGroshong PICC Total =xxx) (N=xxx) (N=xxx) (N=xxx) | | | | | | |
|---|---|---|---|---|---|---|---|---|
| | Power | rPICC | PowerPl | CC SOLO | PowerGros | shong PICC | To | otal |
| | (N=) | xxx) | (N= | xxx) | (N= | xxx) | (N=xxx) | |
| Sherlock TLS used | N | % N % N | | N | % | N | % | |
| missing | | | | | | | | |
| no | | | | | | | | |
| yes | | | | | | | | |
| Overall (non-missing) | | | | | | | | |

| | | | | Type of | Device | | Total<br>(N=xxx)<br>N % | |
|---|---|---|---|---|---|---|---|---|
| | Powe | PowerPICC | | CC SOLO | PowerGros | shong PICC | Total | |
| | (N=) | xxx) | (N= | xxx) | (N= | xxx) | (N=xxx) | |
| Sherlock 3CG used | N | % | N | % | % N % | | N | % |
| missing | | | | | | | | |
| no | | | | | | | | |
| yes | | | | | | | | |
| Overall (non-missing) | | | | | | | | |

| | | | | Type of | Device | | | |
|---|---|---|---|---|---|---|---|---|
| Method used for catheter tip positioning confirmation | Pow | erPICC | PowerPlo | PowerPICC SOLO PowerGroshong PICC | | Total | | |
| | (N: | =xxx) | (N= | xxx) | (N= | xxx) | N % | |
| | N | % | N | % | N | % | N | % |
| missing | | | | | | | | |
| x-ray | | | | | | | | |
| Sherlock 3CG | | | | | | | | |
| Sherlock 3CG+ | | | | | | | | |
| other | | | | | | | | |
| Overall (non-missing) | | | | | | | | |

| | | | | Type of | Device | | | Total<br>(N=xxx)<br>N % |
|---|---|---|---|---|---|---|---|---|
| | Powe | rPICC | PowerPl | CC SOLO | PowerGros | hong PICC | To | otal |
| | (N= | xxx) | (N= | xxx) | (N=xxx) | | (N=xxx) | |
| Stabilization method | N | % | N | % | N | % | N | % |
| missing | | | | | | | | |
| StatLock | | | | | | | | |
| SecurAcath | | | | | | | | |
| Overall (non-missing) | | | | | | | | |

| | | | | Type of | Device | roshong PICC Total N=xxx) (N=xxx) N % | | |
|---|---|---|---|---|---|---|---|---|
| | Power | rPICC | PowerPl | CC SOLO | PowerGros | hong PICC | To | otal |
| | (N=) | (XX) | (N= | xxx) | (N= | xxx) | (N= | (N=xxx) |
| Dressing | N % | | N | % | N | % | N | % |
| missing | | | | | | | | |
| transparent semi-<br>permeable<br>membrane | | | | | | | | |
| gauze | | | | | | | | |
| other | | | | | | | | |
| Overall (non-missing) | | | | | | | | |

| | | | | Type of | Device | | | |
|---|---|---|---|---|---|---|---|---|
| | Powe | PowerPICC | | PowerPICC SOLO | | shong PICC | То | otal |
| | (N= | xxx) | (N=: | xxx) | (N=xxx) | | (N= | xxx) |
| Inserted as per the instructions for use | | | N | % | (N=xxx) (N= | | % | |
| missing | | | | | | | | |
| no | | | | | | | | |
| yes | | | | | | | | |
| Overall (non-missing) | | | | | | | | |

| | | | | Type of | Device | | | |
|---|---|---|---|---|---|---|---|---|
| | Powe | rPICC | PowerPICC SOLO | | PowerGroshong PICC | | Total | |
| | (N= | xxx) | (N= | xxx) | (N=xxx) (N=xxx) | | | xxx) |
| Second implanted line vascular access device present | N | % | N | % | N | % | N | % |
| missing | | | | | | | | |
| no | | | | | | | | |
| yes | | | | | | | | |
| Overall (non-missing) | | | | | | | | |

| | | | | Type of | Device | | | |
|---|---|---|---|---|---|---|---|---|
| | Powe | rPICC | PowerPl | PowerPICC SOLO PowerGroshong PICC | | To | otal | |
| | (N= | xxx) | (N= | xxx) | (N= | xxx) | (N= | xxx) |
| Location of second implanted line | N | % | N | % | N | % | N | % |
| missing | | | | | | | | |
| contralateral | | | | | | | | |
| ipsilateral | | | | | | | | |
| Overall (non-missing) | | | | | | | | |

# **Interim and Final Analysis**


| | | | | Type of | Device | | | |
|---|---|---|---|---|---|---|---|---|
| Type of second device | Power<br>(N=) | | PowerPICC SOLO (N=xxx) | | PowerGroshong PICC (N=xxx) | | Total<br>(N=xxx) | |
| | N | % | N | % | N | % | N | % |
| missing | | | | | | | | |
| subclavian CVC | | | | | | | | |
| IJ CVC | | | | | | | | |
| Overall (non-missing) | | | | | | | | |


• Listing 3.4: Catheter Insertion: Insertion (\*)

Safety Set

**FGK** 

Variables: Type of device, Participant, Catheter length trimmed, Catheter length [cm], External length [cm], Tunneling used, Sherlock TLS used, Sherlock 3CG used, Method to confirm catheter tip positioning / Specification, Stabilization method / Specification, Dressing type / Specification, Inserted as per IFU / Description, Vein lacerated, Vein perforated, Upper arm circumference [cm], Second implanted line present, Location, Type of device / Specification, Comment, Evaluable Set (yes/no)




• Listing 3.5: Participant Location

MDS-19PICCEU01

Safety Set

**Variables:** Type of device, Participant, Sequence No., Participant location / Specification of ward / Specification of other, From / To, Expected maintenance interval for specific location (unit), Expected maintenance interval for dressing change (unit), Expected maintenance interval for catheter insertion site assessment (unit), Device maintained as per site procedure / Description of change, Dressing changed as per site procedure / Description of change, Evaluable Set (yes/no)

#### • Table 3.5: Removal

#### Evaluable Set

| | | Type of Device PowerPICC PowerPICC SOLO PowerGroshong PICC Total (N=xxx) (N=xxx) (N=xxx) (N=xxx) | | | | | | |
|---|---|---|---|---|---|---|---|---|
| | Powe | PowerPICC | | PowerPICC SOLO | | PowerGroshong PICC | | otal |
| | (N= | xxx) | (N= | xxx) | (N= | xxx) | (N= | xxx) |
| Study PICC still in place | N | % | N | % | N | % | N | % |
| missing | | | | | | | | |
| no | | | | | | | | |
| yes | | | | | | | | |
| Overall (non-missing) | | | | | | | | |

| | Type of Device PowerPICC PowerPICC SOLO PowerGroshong PICC Total (N=xxx) (N=xxx) (N=xxx) (N=xxx) N | | | | | | | |
|---|---|---|---|---|---|---|---|---|
| | Powe | rPICC | PowerPl | CC SOLO | PowerGros | hong PICC | To | otal |
| | (N= | xxx) | (N= | xxx) | (N= | xxx) | (N=xxx) | |
| Reason for PICC removal | N % | | N | % | N | % | N | % |
| missing | | | | | | | | |
| therapy completed | | | | | | | | |
| therapy changed or cancelled | | | | | | | | |
| Overall (non-missing) | | | | | | | | |

| | Type of Device | | | | | | | |
|---|---|---|---|---|---|---|---|---|
| | PowerPICC<br>(N=xxx) | | PowerPICC SOLO<br>(N=xxx) | | PowerGroshong PICC (N=xxx) | | Total<br>(N=xxx) | |
| Skin condition around the catheter site normal at removal | N | % | N | % | N | % | N | % |
| missing | 51 | | 75 | | 54 | | 180 | |
| no | 5 | 8.8 | 11 | 15.3 | 0 | 0.0 | 16 | 11.5 |
| yes | 51 | 89.5 | 38 | 52.8 | 7 | 70.0 | 96 | 69.1 |
| unknown | 1 | 1.8 | 23 | 31.9 | 3 | 30.0 | 27 | 19.4 |
| Overall (non-missing) | 57 | 100.0 | 72 | 100.0 | 10 | 100.0 | 139 | 100.0 |

| | Type of Device | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| | PowerPICC<br>(N=xxx) | | | PowerPICC SOLO (N=xxx) | | | Total (N=xxx) | | |
| | No. of Events<br>(N#) | No. of Part.<br>with Event<br>(N) | Part. with<br>Event (%) | No. of Events<br>(N#) | No. of Part.<br>with Event<br>(N) | Part. with<br>Event (%) | No. of Events<br>(N#) | No. of Part.<br>with Event<br>(N) | Part. with<br>Event (%) |
| Specification of abnormal skin condition | | | | | | | | | |
| erythema | | | | | | | | | |
| MARSI | | | | | | | | | |
| Total | | | | | | | | | |

| | | | | | | Type of | Device | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | PowerPICC<br>(N=xxx) | | PowerPICC SOLO<br>(N=xxx) | | | PowerGroshong PICC<br>(N=xxx) | | | Total<br>(N=xxx) | | |
| | No. of<br>Purposes<br>(N#) | No. of<br>Part. with<br>Purpose<br>(N) | Part. with<br>Purpose<br>(%) | No. of<br>Purposes<br>(N#) | No. of<br>Part. with<br>Purpose<br>(N) | Part. with<br>Purpose<br>(%) | No. of<br>Purposes<br>(N#) | No. of<br>Part. with<br>Purpose<br>(N) | Part. with<br>Purpose<br>(%) | No. of<br>Purposes<br>(N#) | No. of<br>Part. with<br>Purpose<br>(N) | Part. with<br>Purpose<br>(%) |
| Use of PICC during the study period | | | | | | | | | | | | |
| pain management | ] | | | | | | | | | | | |
| limited peripheral access | | | | | | | | | | | | |
| Total | | | | | | | | | | | | |

• Listing 3.6: Removal (\*)

Safety Set

**FGK** 

**Variables:** Type of device, Participant, Study PICC still in place, Removal date and time, Reason for removal / Specification of other, Skin condition around the catheter site normal, Specification of abnormal skin condition, Specification of other, Use of PICC line during the study period, Specification of other, Device success, Evaluable Set (yes/no)

• Listing 3.7: Removal: Complications and Performance (\*)

Safety Set

FGK

Variables: Type of device, Participant, PICC always patent, Experience of: Venous thrombosis, Phlebitis, Extravasation, Local infection,

Catheter related bloodstream infection, Evaluable Set (yes/no)

4 Safety

FGK

4.1 Primary Safety Variable

Table 4.1.1: Incidence of Symptomatic Venous Thrombosis (\*)
 Safety Set

| Type of Device | Symptomatic<br>VT | Number of<br>Participants<br>(N) | Participants<br>(%) | Lower 95%<br>Confidence Bound<br>(%) | Upper 95%<br>Confidence Bound<br>(%) |
|---|---|---|---|---|---|
| PowerPICC (N=xxx) | missing | | | | |
| | no | | | | |
| | yes | | | | |
| PowerPICC SOLO (N=xxx) | missing | | | | |
| | no | | | | |
| | yes | | | | |
| PowerGroshong PICC (N=xxx) | missing | | | | |
| | no | | | | |
| | yes | | | | |
| Total (N=xxx) | missing | | | | |
| | no | | | | |
| | yes | | | | |



Statistical Analysis Plan MDS-19PICCEU01

- 4.2 Secondary Safety Variables
- 4.2.1 Complications

• Table 4.2.1.1: Complications (\*)

### Safety Set

| Type of Device | Phlebitis | Number of<br>Participants<br>(N) | Participants (%) | Lower 95%<br>Confidence Bound<br>(%) | Upper 95%<br>Confidence Bound<br>(%) |
|---|---|---|---|---|---|
| PowerPICC (N=xxx) | missing | | | | |
| | no | | | | |
| | yes | | | | |
| PowerPICC SOLO (N=xxx) | missing | | | | |
| | no | | | | |
| | yes | | | | |
| PowerGroshong PICC (N=xxx) | missing | | | | |
| | no | | | | |
| | yes | | | | |
| Total (N=xxx) | missing | | | | |
| | no | | | | |
| | yes | | | | |


| Type of Device | Extravasation | Number of Participants (N) | Participants (%) | Lower 95%<br>Confidence Bound<br>(%) | Upper 95%<br>Confidence Bound<br>(%) |
|---|---|---|---|---|---|
| PowerPICC (N=xxx) | missing | | | | |
| | no | | | | |
| | yes | | | | |
| PowerPICC SOLO (N=xxx) | missing | | | | |
| | no | | | | |
| | yes | | | | |
| PowerGroshong PICC (N=xxx) | missing | | | | |
| | no | | | | |
| | yes | | | | |
| Total (N=xxx) | missing | | | | |
| | no | | | | |
| | yes | | | | |

FGK

| Type of Device | Local Infection* | Number of Participants (N) | Participants (%) | Lower 95%<br>Confidence Bound<br>(%) | Upper 95%<br>Confidence Bound<br>(%) |
|---|---|---|---|---|---|
| PowerPICC (N=xxx) | missing | | | | |
| | no | | | | |
| | yes | | | | |
| PowerPICC SOLO (N=xxx) | missing | | | | |
| | no | | | | |
| | yes | | | | |
| PowerGroshong PICC (N=xxx) | missing | | | | |
| | no | | | | |
| | yes | | | | |
| Total (N=xxx) | missing | | | | |
| | no | | | | |
| | yes | | | | |

**Footnote 1:** \* In total a/b, in PowerPICC c/d, in PowerPICC SOLO e/f, and in PowerGroshong PICC g/h local infections were confirmed according to protocol by presence of pus at the exit site and/or culture confirmed site infection.


| Type of Device | Bloodstream<br>Infection | Number of<br>Participants<br>(N) | Participants (%) | Lower 95%<br>Confidence Bound<br>(%) | Upper 95%<br>Confidence Bound<br>(%) |
|---|---|---|---|---|---|
| PowerPICC (N=xxx) | missing | | | | |
| | no | | | | |
| | yes | | | | |
| PowerPICC SOLO (N=xxx) | missing | | | | |
| | no | | | | |
| | yes | | | | |
| PowerGroshong PICC (N=xxx) | missing | | | | |
| | no | | | | |
| | yes | | | | |
| Total (N=xxx) | missing | | | | |
| | no | | | | |
| | yes | | | | |


| Type of Device | Accidental<br>Dislodgment | Number of<br>Participants<br>(N) | Participants (%) | Lower 95%<br>Confidence Bound<br>(%) | Upper 95%<br>Confidence Bound<br>(%) |
|---|---|---|---|---|---|
| PowerPICC (N=xxx) | missing | | | | |
| | no | | | | |
| | yes | | | | |
| PowerPICC SOLO (N=xxx) | missing | | | | |
| | no | | | | |
| | yes | | | | |
| PowerGroshong PICC (N=xxx) | missing | | | | |
| | no | | | | |
| | yes | | | | |
| Total (N=xxx) | missing | | | | |
| | no | | | | |
| | yes | | | | |

| Type of Device | Vein Laceration | Number of Participants (N) | Participants (%) | Lower 95%<br>Confidence Bound<br>(%) | Upper 95%<br>Confidence Bound<br>(%) |
|---|---|---|---|---|---|
| PowerPICC (N=xxx) | missing | | | | |
| | no | | | | |
| | yes | | | | |
| PowerPICC SOLO (N=xxx) | missing | | | | |
| | no | | | | |
| | yes | | | | |
| PowerGroshong PICC (N=xxx) | missing | | | | |
| | no | | | | |
| | yes | | | | |
| Total (N=xxx) | missing | | | | |
| | no | | | | |
| | yes | | | | |


| Type of Device | Vein Perforation | Number of<br>Participants<br>(N) | Participants (%) | Lower 95%<br>Confidence Bound<br>(%) | Upper 95%<br>Confidence Bound<br>(%) |
|---|---|---|---|---|---|
| PowerPICC (N=xxx) | missing | | | | |
| | no | | | | |
| | yes | | | | |
| PowerPICC SOLO (N=xxx) | missing | | | | |
| | no | | | | |
| | yes | | | | |
| PowerGroshong PICC (N=xxx) | missing | | | | |
| | no | | | | |
| | yes | | | | |
| Total (N=xxx) | missing | | | | |
| | no | | | | |
| | yes | | | | |

- 4.3 Further Safety Variables
- 4.3.1 Adverse Events

• Table 4.3.1.1: Number of Participants with (S)AEs, (S)ADEs, and Related AEs Safety Set

| | | | | | | Type of | Device | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | PowerPICC<br>(N=xxx) | | PowerPICC SOLO<br>(N=xxx) | | | Pow | verGroshong I<br>(N=xxx) | PICC | | Total<br>(N=xxx) | |
| | Number of AEs Number of Part. with AE Part. with | | Number of Part. with AEs AE Part. with | | Number of Part. with AE Part. with AE | | Part. with<br>AE | Number of AEs Number of Part. with AE | | Part. with<br>AE | | |
| | (N#) | (N) | (%) | (N#) | (N) | (%) | (N#) | (N) | (%) | (N#) | (N) | (%) |
| Any AEs | | | | | | | | | | | | |
| Any SAEs | | | | | | | | | | | | |
| Any ADEs | | | | | | | | | | | | |
| Any SADEs | | | | | | | | | | | | |
| Any AEs related to procedure | | | | | | | | | | | | |
| Any AEs related to accessories | | | | | | | | | | | | |



Table 4.3.1.2: AEs by System Organ Class
 Safety Set

| Safety Set | | | | | | | Type of | Device | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | PowerPIC<br>(N=xxx) | С | PowerPICC SOLO<br>(N=xxx) | | | | rGroshong<br>(N=xxx) | PICC | Total<br>(N=xxx) | | |
| | | Number of AEs | Number<br>of Part.<br>with AE | Part. with<br>AE | Number<br>of AEs | Number<br>of Part.<br>with AE | Part.<br>with AE | Number of AEs | Number<br>of Part.<br>with AE | Part.<br>with AE | Number<br>of AEs | Number<br>of Part.<br>with AE | Part.<br>with AE |
| | | (N#) | (N) | (%) | (N#) | (N) | (%) | (N#) | (N) | (%) | (N#) | (N) | (%) |
| System Organ<br>Class (MedDRA) | Preferred Term<br>(MedDRA) | | | | | | | | | | | | |
| Blood and | Anaemia | | | | | | | | | | | | |
| lymphatic system | Thrombocytopenia | | | | | | | | | | | | |
| disorders | Total | | | | | | | | | | | | |
| Candiaa diaandana | Tachycardia | | | | | | | | | | | | |
| Cardiac disorders | Total | | | | | | | | | | | | |
| Total | Total | | | | | | | | | | | | |

Footnote 1: Each participant is counted at most once for the line total. MedDRA version <xx.x> was used for coding.

• Table 4.3.1.3: AEs by System Organ Class and Severity

Safety Set

| | | | | | | | | Type of | Device | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | PowerPICC<br>(N=xxx) | : | Pov | werPICC SO<br>(N=xxx) | LO | Powe | rGroshong<br>(N=xxx) | PICC | | Total<br>(N=xxx) | |
| | | | Number of AEs | Number<br>of Part.<br>with AE | Part. with AE | Number of AEs | Number<br>of Part.<br>with AE | Part.<br>with AE | Number of AEs | Number<br>of Part.<br>with AE | Part.<br>with AE | Number of AEs | Number<br>of Part.<br>with AE | Part.<br>with AE |
| | | | (N#) | (N) | (%) | (N#) | (N) | (%) | (N#) | (N) | (%) | (N#) | (N) | (%) |
| System<br>Organ Class<br>(MedDRA) | Preferred Term<br>(MedDRA) | Severity | | | | | | | | | | | | |
| | | mild | | | | | | | | | | | | |
| | Anaemia | moderate | | | | | | | | | | | | |
| | severe | | | | | | | | | | | | | |
| Blood and | | mild | | | | | | | | | | | | |
| lymphatic<br>system | Thrombocytopenia | moderate | | | | | | | | | | | | |
| disorders | | severe | | | | | | | | | | | | |
| | | mild | | | | | | | | | | | | |
| | Total | moderate | | | | | | | | | | | | |
| | | severe | | | | | | | | | | | | |
| | | mild | | | | | | | | | | | | |
| Total | Total | moderate | | | | | | | | | | | | |
| | | severe | | | | | | | | | | | | |

• Table 4.3.1.4: Serious AEs by System Organ Class

Safety Set

FGK

Note: The same table layout as used for table AEs by system organ class will be used. Only serious AEs will be tabulated.

Footnote 1: Adverse events documented as serious on the AE form are tabulated.

• Table 4.3.1.5: Non-serious AEs by System Organ Class

Safety Set

*Note:* The same table layout as used for table AEs by system organ class will be used. Only non-serious AEs will be tabulated.

Footnote 1: Adverse events documented as non-serious on the AE form are tabulated.

• Table 4.3.1.6: Adverse Device Effects by System Organ Class

Safety Set

**FGK** 

Note: The same table layout as used for table AEs by system organ class will be used.

Footnote 1: Adverse events documented as related to device on the AE form are tabulated.

- Table 4.3.1.7: Serious Adverse Device Effects by System Organ Class
  - Safety Set

Note: The same table layout as used for table AEs by system organ class will be used. Only serious AEs will be tabulated.

- Footnote 1: Serious adverse events documented as related to device on the AE form are tabulated.
- Footnote 2: Each participant is counted at most once for the line total. MedDRA version <xx.x> was used for coding.

• Table 4.3.1.8: AEs Related to Procedure by System Organ Class

Safety Set

**Note:** The same table layout as used for table AEs by system organ class will be used. Only AEs related to procedure will be tabulated.

Footnote 1: Adverse events documented as related to procedure on the AE form are tabulated.

• Table 4.3.1.9: AEs Related to Accessories by System Organ Class

Safety Set

Note: The same table layout as used for table AEs by system organ class will be used. Only AEs related to Accessories will be tabulated.

Footnote 1: Adverse events documented as related to accessories on the AE form are tabulated.

• Listing 4.3.1.1: Adverse Events (\*)

Safety Set

Variables: Type of device, Participant + all variables on AE-form + Preferred term and system organ class, Study day of AE, Duration of AE,

Evaluable Set (yes/no)

• Listing 4.3.1.2: Serious Adverse Events - AE Form

Safety Set

**Variables:** Type of device, Participant + all variables on AE-form + Preferred term and system organ class, Study day of AE, Duration of AE, Evaluable Set (yes/no)

Footnote 1: Adverse events documented as serious on the AE form are listed only.

• Listing 4.3.1.3: Serious Adverse Events - SAE Form

Safety Set

Variables: Type of device, Participant + all variables on SAE-form as entered by the investigator, Evaluable Set (yes/no)

4.3.2 Device Deficiencies

• Listing 4.3.2.1: Device Deficiencies

Safety Set

FGK

Variables: Type of Device, Participant + all variables on device deficiency-form, Evaluable Set (yes/no)



- 5 Performance Analysis
- 5.1 Analysis of Primary Performance Variable

**Interim and Final Analysis** 

FGK

• Table 5.1.1: PICCs that remain in place through completion of therapy (\*) Evaluable Set

| Type of Device | PICCs that remain in place<br>through completion of<br>therapy | Number of<br>Participants<br>(N) | Participants (%) | Lower 95%<br>Confidence Bound<br>(%) | Upper 95%<br>Confidence Bound<br>(%) |
|---|---|---|---|---|---|
| PowerPICC (N=xxx) | missing | | | | |
| | no | | | | |
| | yes | | | | |
| PowerPICC SOLO (N=xxx) | missing | | | | |
| | no | | | | |
| | yes | | | | |
| PowerGroshong PICC (N=xxx) | missing | | | | |
| | no | | | | |
| | yes | | | | |
| Total (N=xxx) | missing | | | | |
| | no | | | | |
| | yes | | | | |

**5.2** Analysis of Secondary Performance Variables

• Table 5.2.1: Patent Catheters (\*)

### Evaluable Set

| Type of Device | Patent<br>Catheter | Number of<br>Catheters (N) | Catheters (%) | Lower 95%<br>Confidence Bound<br>(%) | Upper 95%<br>Confidence Bound<br>(%) |
|---|---|---|---|---|---|
| PowerPICC (N=xxx) | missing | | | | |
| | no | | | | |
| | yes | | | | |
| PowerPICC SOLO (N=xxx) | missing | | | | |
| | no | | | | |
| | yes | | | | |
| PowerGroshong PICC (N=xxx) | missing | | | | |
| | no | | | | |
| | yes | | | | |
| Total (N=xxx) | missing | | | | |
| | no | | | | |
| | yes | | | | |

• Table 5.2.2: Placement Success in Single Insertion Attempt (\*)

Safety Set

| Type of Device | Placement Success in a Single Insertion Attempt | Number of<br>Catheters (N) | Catheters (%) | Lower 95%<br>Confidence Bound<br>(%) | Upper 95%<br>Confidence Bound<br>(%) |
|---|---|---|---|---|---|
| PowerPICC (N=xxx) | missing | | | | |
| | no | | | | |
| | yes | | | | |
| PowerPICC SOLO (N=xxx) | missing | | | | |
| | no | | | | |
| | yes | | | | |
| PowerGroshong PICC (N=xxx) | missing | | | | |
| | no | | | | |
| | yes | | | | |
| Total (N=xxx) | missing | | | | |
| | no | | | | |
| | yes | | | | |

• Table 5.2.3: Usability: Ease of Insertion – Guidewire (\*)

Safety Set

| | Type of Device | | | | | | | |
|---|---|---|---|---|---|---|---|---|
| Difficulty to use the guidewire | PowerPICC<br>(N=xxx) | | PowerPICC SOLO (N=xxx) | | PowerGroshong PICC (N=xxx) | | Total<br>(N=xxx) | |
| | N | % | N | % | N | % | N | % |
| missing | | | | | | | | |
| very difficult | | | | | | | | |
| difficult | | | | | | | | |
| Overall (non-missing) | | | | | | | | |

| | Type of Device | | | | | | | |
|---|---|---|---|---|---|---|---|---|
| | PowerPICC | | PowerPICC SOLO | | PowerGroshong PICC | | То | otal |
| | (N= | xxx) | (N= | xxx) | (N=xxx) | | (N=xxx) | |
| Force to advance the guidewire acceptable | N | % | N | % | N | % | N | % |
| missing | | | | | | | | |
| no | | | | | | | | |
| yes | | | | | | | | |
| Overall (non-missing) | | | | | | | | |

| | Type of Device | | | | | | | |
|---|---|---|---|---|---|---|---|---|
| | PowerPICC | | PowerPl | CC SOLO | PowerGroshong PICC | | Total | |
| | (N= | xxx) | (N= | xxx) | (N=xxx) | | (N=xxx) | |
| Difficulty to withdraw/remove the guidewire | N | % | N | % | N | % | N | % |
| missing | | | | | | | | |
| very difficult | | | | | | | | |
| difficult | | | | | | | | |
| Overall (non-missing) | | | | | | | | |

| | Type of Device | | | | | | | |
|---|---|---|---|---|---|---|---|---|
| Force to withdraw/remove the guidewire acceptable | PowerPICC<br>(N=xxx) | | PowerPICC SOLO (N=xxx) | | PowerGroshong PICC (N=xxx) | | Total<br>(N=xxx) | |
| | N | % | N | % | N | % | N | % |
| missing | | | | | | | | |
| no | | | | | | | | |
| yes | | | | | | | | |
| Overall (non-missing) | | | | | | | | |

| | Type of Device | | | | | | |
|---|---|---|---|---|---|---|---|
| | PowerPICC<br>(N=xxx) | | PowerPICC SOLO (N=xxx) | | PowerGroshong PICC<br>(N=xxx) | | Total<br>(N=xxx) |
| Agreement on Integrity | N | % | N | N % N % | | N | % |
| missing | | | | | | | |
| strongly disagree | | | | | | | |
| disagree | | | | | | | |
| Overall (non-missing) | | | | | | | |

| | Type of Device | | | | | | | |
|---|---|---|---|---|---|---|---|---|
| | Powe | PowerPICC | | PowerPICC SOLO | | PowerGroshong PICC | | otal |
| Agreement on Guidewire facilitated placement | (N=xxx) | | (N=xxx) | | (N=xxx) | | (N=xxx) | |
| | N | % | N | % | N | % | N | % |
| missing | | | | | | | | |
| strongly disagree | | | | | | | | |
| disagree | | | | | | | | |
| Overall (non-missing) | | | | | | | | |
Table 5.2.4: Usability: Ease of Insertion – Guidewire – Basic Statistics (\*)
 Safety Set

| | | | Type of Device | | Total |
|---|---|---|---|---|---|
| | | PowerPICC<br>(N=xxx) | PowerPICC SOLO (N=xxx) | PowerGroshong PICC (N=xxx) | (N=xxx) |
| | N | | | | |
| | missing | | | | |
| | mean | | | | |
| Difficulty to | SD | | | | |
| use the | minimum | | | | |
| guidewire | 1st quartile | | | | |
| | median | | | | |
| | 3rd quartile | | | | |
| | maximum | | | | |

| | | | Type of Device | | Total |
|---|---|---|---|---|---|
| | | PowerPICC<br>(N=xxx) | PowerPICC SOLO (N=xxx) | PowerGroshong PICC (N=xxx) | (N=xxx) |
| | N | | | | |
| | missing | | | | |
| | mean | | | | |
| Difficulty to | SD | | | | |
| withdraw/remove | minimum | | | | |
| the guidewire | 1st quartile | | | | |
| | median | | | | |
| | 3rd quartile | | | | |
| | maximum | | | | |

| | | | Type of Device | | Total |
|---|---|---|---|---|---|
| | | PowerPICC<br>(N=xxx) | PowerPICC SOLO (N=xxx) | · | |
| | N | | | | |
| | missing | | | | |
| | mean | | | | |
| | SD | | | | |
| Agreement on Integrity | minimum | | | | |
| ······································ | 1st quartile | | | | |
| | median | | | | |
| | 3rd quartile | | | | |
| | maximum | | | | |

| | | | Type of Device | | Total |
|---|---|---|---|---|---|
| | | PowerPICC<br>(N=xxx) | PowerPICC SOLO (N=xxx) | PowerGroshong PICC (N=xxx) | (N=xxx) |
| | N | | | | |
| | missing | | | | |
| | mean | | | | |
| Agreement | SD | | | | |
| on Guidewire facilitated | minimum | | | | |
| placement | 1st quartile | | | | |
| | median | | | | |
| | 3rd quartile | | | | |
| | maximum | | | | |

• Table 5.2.5: Usability: Ease of Insertion – Stylet (\*)

Safety Set

| | | Type of Device | | | | | | |
|---|---|---|---|---|---|---|---|---|
| | PowerPICC<br>(N=xxx) | | PowerPICC SOLO (N=xxx) | | PowerGros | shong PICC | Total | |
| | | | | | (N=xxx) | | (N=xxx) | |
| Difficulty to use the stylet | N | % | N | % | N | % | N | % |
| missing | | | | | | | | |
| 1 = very difficult | | | | | | | | |
| 2 = difficult | | | | | | | | |
| Overall (non-missing) | | | | | | | | |

| | | Type of Device | | | | | | |
|---|---|---|---|---|---|---|---|---|
| | PowerPICC<br>(N=xxx) | | PowerPl | CC SOLO | PowerGros | shong PICC | То | otal |
| | | | (N=xxx) | | (N=xxx) | | (N=xxx) | |
| Force to advance the stylet/catheter acceptable | N | % | N | % | N | % | N | % |
| missing | | | | | | | | |
| no | | | | | | | | |
| yes | | | | | | | | |
| Overall (non-missing) | | | | | | | | |

| | | Type of Device | | | | | | |
|---|---|---|---|---|---|---|---|---|
| | PowerPICC<br>(N=xxx) | | PowerPl | CC SOLO | PowerGros | shong PICC | Total | |
| | | | (N=xxx) | | (N=xxx) | | (N=xxx) | |
| Difficulty to withdraw/remove the stylet/catheter | N | % | N | % | N | % | N | % |
| missing | | | | | | | | |
| 1 = very difficult | | | | | | | | |
| 2 = difficult | | | | | | | | |
| Overall (non-missing) | | | | | | | | |

| Force to withdraw/remove the guidewire acceptable | Type of Device | | | | | | | |
|---|---|---|---|---|---|---|---|---|
| | PowerPICC<br>(N=xxx) | | PowerPICC SOLO<br>(N=xxx) | | PowerGroshong PICC (N=xxx) | | Total<br>(N=xxx) | |
| | N | % | N | % | N | % | N | % |
| missing | | | | | | | | |
| no | | | | | | | | |
| yes | | | | | | | | |
| Overall (non-missing) | | | | | | | | |

| | | Type of Device | | | | | |
|---|---|---|---|---|---|---|---|
| | PowerPICC<br>(N=xxx) | | | CC SOLO | | shong PICC | Total |
| | | | (N=xxx) | | (N=xxx) | | (N=xxx) |
| Agreement on Integrity | | | | | | | |
| missing | | | | | | | |
| no | | | | | | | |
| yes | | | | | | | |
| Overall (non-missing) | | | | | | | |

| | | Type of Device | | | | | | |
|---|---|---|---|---|---|---|---|---|
| | Powe | PowerPICC | | CC SOLO | PowerGros | shong PICC | To | otal |
| | (N=xxx) | | (N=xxx) | | (N=xxx) | | (N=xxx) | |
| Stylet/catheter facilitated placement | N | % | N | % | N | % | N | % |
| missing | | | | | | | | |
| 1 = strongly disagree | | | | | | | | |
| 2 = disagree | | | | | | | | |
| Overall (non-missing) | | | | | | | | |

| | | Type of Device | | | | | | |
|---|---|---|---|---|---|---|---|---|
| Sherlock 3CG Pre-Loaded question answered | PowerPICC<br>(N=xxx) | | PowerPl | CC SOLO | PowerGros | shong PICC | Total | |
| | | | (N=xxx) | | (N=xxx) | | (N=xxx) | |
| | N | % | N | % | N | % | N | % |
| missing | | | | | | | | |
| yes | | | | | | | | |
| not applicable / not used | | | | | | | | |
| Overall (non-missing) | | | | | | | | |

| | | Type of Device | | | | | | |
|---|---|---|---|---|---|---|---|---|
| | Powe | PowerPICC | | PowerPICC SOLO | | shong PICC | Total | |
| | (N=xxx) | | (N=xxx) | | (N=xxx) | | (N=xxx) | |
| Sherlock 3CG Pre-Loaded stylet aided | N | % | N | % | N | % | N | % |
| missing | | | | | | | | |
| 1 = strongly disagree | | | | | | | | |
| 2 = disagree | | | | | | | | |
| Overall (non-missing) | | | | | | | | |

| | Type of Device | | | | | | | |
|---|---|---|---|---|---|---|---|---|
| , | PowerPICC | | PowerPICC SOLO | | PowerGroshong PICC | | Total<br>(N=xxx) | |
| | (N=: | xxx) | (N=xxx) (N=xxx) | | | | | |
| Sherlock Tip Location System (TLS) Pre-Loaded stylet question answered | N | % | N | % | N | % | N | % |
| missing | | | | | | | | |
| yes | | | | | | | | |
| not applicable / not used | | | | | | | | |
| Overall (non-missing) | | | | | | | | |

| | Type of Device | | | | | | | |
|---|---|---|---|---|---|---|---|---|
| | PowerPICC<br>(N=xxx) | | | | PowerGroshong PICC | | Total | |
| | | | | | =xxx) (N | | =xxx) | |
| Sherlock Tip Location System (TLS) Pre-Loaded stylet aided | N | % | N | % | N | % | N | % |
| missing | | | | | | | | |
| 1 = strongly disagree | | | | | | | | |
| 2 = disagree | | | | | | | | |
| Overall (non-missing) | | | | | | | | |

Table 5.2.6: Usability: Ease of Insertion – Stylet – Basic Statistics (\*)
 Safety Set

| | | Type of Device | | |
|---|---|---|---|---|
| | | PowerPICC<br>(N=xxx) | PowerPICC SOLO (N=xxx) | Total<br>(N=xxx) |
| | N | | | |
| | missing | | | |
| | mean | | | |
| | SD | | | |
| Difficulty to use the stylet | minimum | | | |
| | 1st quartile | | | |
| | median | | | |
| | 3rd quartile | | | |
| | maximum | | | |

| | | Type of Device | | | Total |
|---|---|---|---|---|---|
| | | PowerPICC<br>(N=xxx) | PowerPICC SOLO (N=xxx) | PowerGroshong PICC (N=xxx) | (N=xxx) |
| | N | | | | |
| | missing | | | | |
| | mean | | | | |
| Difficulty to | SD | | | | |
| withdraw/remove the | minimum | | | | |
| stylet/catheter | 1st quartile | | | | |
| | median | | | | |
| | 3rd quartile | | | | |
| | maximum | <u> </u> | | | · |

| | | | Total | | |
|---|---|---|---|---|---|
| | | PowerPICC<br>(N=xxx) | PowerPICC SOLO (N=xxx) | PowerGroshong PICC (N=xxx) | (N=xxx) |
| | N | | | | |
| | missing | | | | |
| | mean | | | | |
| Agreement on | SD | | | | |
| stylet/catheter facilitated | minimum | | | | |
| placement | 1st quartile | | | | |
| | median | | | | |
| | 3rd quartile | | | | |
| | maximum | | | | |

| | | | Total | | |
|---|---|---|---|---|---|
| | | PowerPICC<br>(N=xxx) | PowerPICC SOLO (N=xxx) | PowerGroshong PICC (N=xxx) | (N=xxx) |
| | N | | | | |
| | missing | | | | • |
| | mean | | | | |
| Sherlock | SD | | | | |
| 3CG Pre-<br>Loaded | minimum | | | | |
| Stylet aided | 1st quartile | | | | |
| | median | | | | |
| | 3rd quartile | | | | |
| | maximum | | | | |

## **Interim and Final Analysis**


| | | | Total | | |
|---|---|---|---|---|---|
| | | PowerPICC<br>(N=xxx) | PowerPICC SOLO (N=xxx) | PowerGroshong PICC (N=xxx) | (N=xxx) |
| | N | | | | |
| | missing | | | | |
| | mean | | | | |
| Sherlock Tip<br>Location | SD | | | | |
| System (TLS) | minimum | | | | |
| Pre-Loaded<br>Stylet aided | 1st quartile | | | | |
| • | median | | | | |
| | 3rd quartile | | | | |
| | maximum | | | | |

## **Interim and Final Analysis**

Appendix A


• Listing 5.2.1: Usability: Ease of Insertion – Guidewire (\*)

Safety Set

**Variables:** Type of device, Participant, Difficulty to use the guidewire / Explanation, Force acceptable to advance the guidewire / Explanation, Difficulty to withdraw/remove the guidewire / Explanation, Force to withdraw/remove the guidewire acceptable / Explanation, Agreement on: Integrity / Explanation, Guidewire facilitated placement / Explanation, Evaluable Set (yes/no)

**Note:** Type of devices will be displayed as "by-variable" within a subtitle.

## **Interim and Final Analysis**

Appendix A


• Listing 5.2.2: Usability: Ease of Insertion – Stylet (\*)

Safety Set

Variables: Type of device, Participant, Difficulty to use the stylet / Explanation, Force to advance the stylet/catheter acceptable / Explanation, Difficulty to withdraw/remove the stylet/catheter / Explanation, Force to withdraw/remove the stylet/catheter acceptable / Explanation, Agreement on: Integrity / Explanation, Stylet/catheter facilitated placement / Explanation, Sherlock 3CG Pre-Loaded Stylet aided / Explanation, Sherlock Tip Location System (TLS) Pre-Loaded Stylet aided / Explanation

Note: Type of devices will be displayed as "by-variable" within a subtitle.


6 Protocol Deviations


• Listing 6.1: Protocol Deviations (eCRF)

**Enrolled Set** 

*Variables:* Type of Device, Participant, Sequence No., Category (including specification of other), Date of deviation, Description, Action / outcome, Evaluable Set (yes/no)

**Note:** Type of devices will be displayed as "by-variable" within a subtitle.